CLINICAL TRIAL: NCT00611065
Title: Imaging of Prostate Cancer Using Two-dimensional MR Spectroscopy and Diffusion Tensor Imaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no funding to proceed.
Sponsor: University of California, Irvine (Other)
Responsible Party: Min-Ying Su, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCI-HS-2007-5671
Record Dates: First submitted 2008-01-12; First posted 2008-02-08 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Prostate Lesions
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: magnetic resonance imaging — MR contrast agent (0.1 mmol/kg)

SUMMARY:
The goal is to develop MR imaging techniques to improve delineation of cancer extent, and to improve differential diagnosis between prostate cancer and benign prostate hyperplasia or other benign diseases.

ELIGIBILITY:
Inclusion Criteria:

1. A male older than 21 years of age and under age of 80,
2. Either a normal healthy volunteer; a patient who has confirmed prostate cancer and decided to receive prostatectomy; or a patient who has persistent elevated PSA higher than 4.0 ng/ml, and with a prior benign biopsy scheduled to receive the second biopsy.

Exclusion Criteria:

1. Unwilling to give informed consent,
2. Have implanted prosthetic heart valves, pacemaker, neuro-stimulation devices, surgical clips (hemostatic clips) or other metallic implants,
3. Have engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or have imbedded metal fragments from military activities,
4. Have received orthodontic work involving ferromagnetic materials,
5. Claustrophobic,
6. Unable to lie down still for 60 minutes.

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that multi-voxel MR spectroscopy and diffusion tensor imaging can accurately diagnose prostate cancer and benign diseases, also to provide an accurate disease extent. | at completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Min-Ying Su, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Center for Functional Onco-Imaging, University of California, Irvine, California, United States